CLINICAL TRIAL: NCT00250926
Title: A Phase II Study of the Combination Bortezomib (Velcade, PS-341), Dexamethasone, and Rituximab in Patients With Waldenstroms Macroglobulinemia
Brief Title: Study of the Combination of Bortezomib, Dexamethasone, and Rituximab in Patients With Waldenstroms Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Steven P. Treon, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-180
Record Dates: First submitted 2005-11-08; First posted 2005-11-09 (Estimated); Results first posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: bortezomib; dexamethasone; rituximab
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib, Dexamethasone, Rituximab (Experimental): A cycle of therapy consisted of bortezomib 1.3 mg/m(2) intravenously; dexamethasone 40 mg on days 1, 4, 8, and 11; and rituximab 375 mg/m(2) on day 11. Patients received four consecutive cycles for induction therapy and then four more cycles, each given 3 months apart, for maintenance therapy.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Rituximab

INTERVENTIONS:
Drug: Bortezomib — Given intravenously on days 1, 4, 8, and 11 of a 21-day cycle for 8 cycles
  Other Names: Bortezomib (Velcade)
Drug: Dexamethasone — Given intravenously on days 1, 4, 8, and 11 of a 21-day cycle for 8 cycles
  Other Names: Dexamethasone (Decadron)
Drug: Rituximab — Given intravenously after bortezomib and dexamethasone on day 11 of a 21-day cycle for 8 cycles
  Other Names: Rituximab (Rituxan)

SUMMARY:
The purpose of this study is to find out if the combination of bortezomib (Velcade), dexamethasone (Decadron) and rituximab (Rituxan) is effective in treating Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
* This is an open-label study which means both the patient and the doctor will know what drugs and doses the patient is receiving throughout the study.
* Patients will receive 8 cycles of study treatment with bortezomib, dexamethasone and rituximab. Each cycle is 21 days long. Therapy is given on the first, fourth, eighth and eleventh day of each cycle, followed by a 10 day rest period. The first 4 cycles will be given one after the other. Three months after completing the fourth cycle of therapy, patients will receive one cycle of therapy every three months for a total of four more cycles.
* On the first, fourth, eighth and eleventh day of each cycle, the patient will receive bortezomib and dexamethasone as an intravenous injection through a needle in your vein. On the eleventh day only, the patient will also receive rituximab as an intravenous infusion after getting bortezomib and dexamethasone.
* Prior to each infusion of rituximab therapy, the patient will be asked to take some medications to prevent or reduce side effects of rituximab. These medications are benadryl, tylenol, and possibly more steroids. The doctor will determine which of these drugs are appropriate for the individual patient.
* During the rituximab infusion, the patients blood pressure and pulse will be monitored frequently and the infusion rate may be decreased depending upon the side effects experienced.
* After therapy is completed, the patient will be followed every three months for 2 more years for office visits and laboratory tests to determine how well they are doing and if the therapy continues to benefit them.

ELIGIBILITY:
Inclusion Criteria:

* Clinicopathological diagnosis of Waldenstrom's macroglobulinemia (WM)
* No previous therapy for WM
* Measurable disease, defined as presence of immunoglobulin M (IgM) paraprotein with a minimum IgM level of greater than or equal to 2 times the upper limit of each institution's normal value
* CD20 positive disease based on any previous bone marrow immuno-histochemistry or flow cytometric analysis performed up to 3 months prior to enrollment
* Karnofsky performance status > 60
* Life expectancy > 3 months
* AST (SGOT) < 3 x ULN
* ALT (SGPT) < 3 x ULN
* Total bilirubin < 2 x ULN
* Calculated or measured creatinine clearance > 30mL/minute
* Serum sodium > 130 mmol/L
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control
* Male subject agrees to use an acceptable method for contraception for the duration of the study

Exclusion Criteria:

* Previous therapy for Waldenstrom's macroglobulinemia
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Hypersensitivity to dexamethasone, boron or mannitol
* Pregnant or breast-feeding women
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-10; Primary Completion 2007-03 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P. Treon, MD, MA, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Result] Treon SP, Ioakimidis L, Soumerai JD, Patterson CJ, Sheehy P, Nelson M, Willen M, Matous J, Mattern J 2nd, Diener JG, Keogh GP, Myers TJ, Boral A, Birner A, Esseltine DL, Ghobrial IM. Primary therapy of Waldenstrom macroglobulinemia with bortezomib, dexamethasone, and rituximab: WMCTG clinical trial 05-180. J Clin Oncol. 2009 Aug 10;27(23):3830-5. doi: 10.1200/JCO.2008.20.4677. Epub 2009 Jun 8. PMID 19506160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient clinic at DFCI
Pre-assignment Details: Symptomatic patients with Waldenstrom's requiring therapy, previously untreated.
Period: Overall Study
Arm/Group | Bortezomib, Dexamethasone, Rituximab
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: This outcome measure was to assess the safety and tolerability of bortezomib, dexamethasone and rituximab in patients with untreated Waldenstroms macroglobulinemia.
Time Frame: 33.2 months
Population: All enrolled patients
Measure: Number; unit: participants
Arm/Group | Bortezomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 23
participants | 23

2. Primary Outcome: Response Rate
Description: This outcome measure was to determine the response rate along with attainment of stable disease and time to disease progression following treatment with this patient population. The response rates were defined as follows.
  A complete response (CR) was defined as having resolution of all symptoms, normalization of serum IgM levels with complete disappearance of IgM paraprotein by immunofixation, absence of bone marrow disease by bone marrow biopsy and aspiration, and resolution of any adenopathy or splenomegaly. A near complete response (nCR) was defined as fulfilling all CR criteria in the presence of a positive immunofixation study. Patients with very good partial response (VGPR), partial response (PR), and minor response (MR) were defined as having a ≥ 90%, ≥ 50%, and 25% to 49% reduction in serum IgM levels, respectively. Progressive disease (PD) occurred when a more than 25% increase in serum IgM level or progression of clinically significant disease parameters was observed.
Time Frame: 33.2 months
Population: all enrolled patients
Measure: Number; unit: participants
Arm/Group | Bortezomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 23
participants
  Complete Response (CR) | 3
  Near Complete Response (nCR) | 2
  Very Good Partial Response (VGPR) | 3
  Partial Response (PR) | 11
  Minor Response (MR) | 3
  Stable Disease | 1

3. Primary Outcome: Time to Best Response
Time Frame: 33.2 months
Measure: Median (Full Range); unit: Months
Arm/Group | Bortezomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 23
Months | 15 [0.7 to 26]

4. Primary Outcome: Time to Progression
Description: Progressive Disease (PD) will be defined as a greater than 25% increase in serum IgM monoclonal protein levels from the lowest attained response value as determined by serum electrophoresis, confirmed by at least one other investigation, or progression of clinically significant disease related symptom(s).
Time Frame: 42 months
Population: The median time to progression was not achieved as follow-up ended before half the participants had a PD event.
Measure: Median (Full Range); unit: months
Arm/Group | Bortezomib, Dexamethasone, Rituximab
Number analyzed (Participants) | 23
months | NA [6 to NA] — The median time to progression was not met before the follow-up time for the protocol was complete. Most patients had not had a PD event at the 42 month cut-off.

ADVERSE EVENTS:
Arm/Group | Bortezomib, Dexamethasone, Rituximab
Serious Adverse Events (participants affected / at risk) | 19/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib, Dexamethasone, Rituximab (N=23)
Peripheral Neuropathy (Nervous system disorders) | 7 (7) — 7 patients, grade 3
Neutropenia (Blood and lymphatic system disorders) | 6 (6) — 6 patients, grade 3
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) — 2 patients, grade 3
myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) — 1 patient, grade 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 1 patient, grade 3
Infection with Neutropenia (Blood and lymphatic system disorders) | 1 (1) — 1 patient, grade 3
hypotension (General disorders) | 1 (1) — 1 patient, grade 3
arrythmia (Cardiac disorders) | 1 (1) — 1 patient, grade 3
anemia (Blood and lymphatic system disorders) | 1 (1) — 1 patient, grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib, Dexamethasone, Rituximab (N=23)
Peripheral Neuropathy (Nervous system disorders) | 9 (9) — 9 patients, grade 2
Infection without Neutropenia (Infections and infestations) | 10 (10) — 10 patients, grade 2
Anemia (Blood and lymphatic system disorders) | 18 (18) — 18 patients, grade 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) — 8 patients, grade 2
neutropenia (Cardiac disorders) | 6 (6) — 6 patients, grade 2
hyeprglycemia (Endocrine disorders) | 6 (6) — 6 patients, grade 2
herpes zoster (Infections and infestations) | 5 (5) — 5 patients, grade 2.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — 2 patients, grade 2
Fatigue (General disorders) | 4 (4) — 4 patients, grade 2
Insomnia (General disorders) | 3 (3) — 3 patients, grade 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) — 3 patients, grade 2
dehydration (General disorders) | 3 (3) — 3 patients, grade 2
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) — 3 patients, grade 2
arrythmia (Cardiac disorders) | 2 (2) — 2 patients, grade 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No